CLINICAL TRIAL: NCT05187871
Title: Establishment and Research for Rapid Diagnosis of Postoperative Abdominal Infection Based on Metagenomic Sequencing
Brief Title: Study for Rapid Diagnosis of Postoperative Abdominal Infection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRDPAI
Record Dates: First submitted 2021-12-08; First posted 2022-01-12 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2021-11

CONDITIONS: Postoperative Infection; Abdominal Surgery; Intra-abdominal Infection; Postoperative Fever
MeSH Terms: conditions — Intraabdominal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective and exploratory study, which utilizes non-targeted metagenomic next-generation sequencing (mNGS) detecting drain fluid from patients who are suspected of postoperative abdominal infection. This study aims to explore the clinical value of mNGS in the rapid diagnosis of postoperative abdominal infection, to refine the pathogenic bacteria spectrum, and to establish a novel procedure for postoperative abdominal infection diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who receive abdominal operations with routinely abdominal drainage placement.
2. Abdominal infection is suspected by the clinicians, and one of the following conditions is met:

   1. Temperature ≥38℃;
   2. One of the following laboratory indicators: WBC≥10×10^9/L, PCT≥0.5ng/ml, hsCRP≥100mg/L.

Exclusion Criteria:

1. Patients who are diagnosed with the abdominal infection before surgery.
2. Evidence of non-abdominal infection is clear and could explain the clinical symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receive abdominal surgery including pancreatic, gastrointestinal, biliary surgery, etc. with routinely placing abdominal drainage in Peking Union Medical College Hospital. They are clinically suspected with postoperative abdominal infection.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The pathogenic spectrum of postoperative abdominal infection | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Consistency between mNGS and conventional culture methods | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhu R, Hong X, Zhang D, Xiao Y, Xu Q, Wu B, Guo J, Han X, Yang Q, Zhao Y, Wu W. Application of metagenomic sequencing of drainage fluid in rapid and accurate diagnosis of postoperative intra-abdominal infection: a diagnostic study. Int J Surg. 2023 Sep 1;109(9):2624-2630. doi: 10.1097/JS9.0000000000000500. PMID 37288562